CLINICAL TRIAL: NCT03516565
Title: Modulation of Matrix Metalloproteinases-8, -9 and Endogenous Tissue Inhibitor-1 in Oral Biofluids During Pregnancy and Postpartum
Brief Title: Matrix Metalloproteinases's in Oral Biofluids During Pregnancy and Postpartum
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Veli Özgen Öztürk, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: BAP-18
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy
Keywords: gingivitis; saliva; gingival crevicular fluid
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnancy group: Pregnant group included women, who were in their second trimester (weeks 16-24) and third trimester (weeks 25-34)
  Interventions: Other: Saliva collection; Other: GCF collection
- Postpartum group: Postpartum group included women, who were evaluated 6 months after giving birth
  Interventions: Other: Saliva collection; Other: GCF collection
- Non-pregnant group: Women who were systemically healthy and non-pregnant.
  Interventions: Other: Saliva collection; Other: GCF collection

INTERVENTIONS:
Other: Saliva collection
Other: GCF collection

SUMMARY:
The aim of this study was to investigate salivary and gingival crevicular fluid (GCF) levels of MMP-8, MMP-9 and TIMP-1 during 2/3 trimester of pregnancy and after delivery

DETAILED DESCRIPTION:
MMP-8 and MMP-9 have been reported to reflect the inflammatory status in periodontal tissues and, therefore represent as potential biomarkers of periodontitis. The balance between tissue inhibitors of metalloproteinases (TIMPs) and MMPs play an important role in maintaining the integrity of healthy periodontium.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant group included women, who were in their second trimester (weeks 16-24) and third trimester (weeks 25-34)

Exclusion Criteria:

* (a) any known systemic disease, (b) periodontal treatment within the last six months, (c) patients having less than 10 teeth, (d) smokers and (e) individuals with BMI > 30 kg/m2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women were systemically healthy
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Changing MMP-8 levels | 6 months
  Salivary and GCF level measured by IFMA
Changing MMP-9 levels | 6 months
  Salivary and GCF level measured by ELISA
Changing TIMP-1 levels | 6 months
  Salivary and GCF level measured by ELISA

IPD SHARING:
Plan to Share IPD: No